CLINICAL TRIAL: NCT00459901
Title: Phase II Trial of OSI-774 (Erlotinib, Tarceva™,) and Capecitabine for Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Study of the Antitumor Activity of Capecitabine in Combination With Erlotinib in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted by drug manufacturer
Sponsor: Peter Kozuch (Other)
Collaborators: Hoffmann-La Roche (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Peter Kozuch, Attending, Beth Israel Medical Center
Organization: Beth Israel Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022-03; XEL308
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Erlotinib Hydrochloride; Capecitabine

INTERVENTIONS:
Drug: Erlotinib and capecitabine

SUMMARY:
To document the antitumor activity of capecitabine in combination with erlotinib in patients with previously untreated metastatic colorectal cancer. Time to tumor progression, objective response rate, time to confirmed response rate, duration of confirmed response rate, time to treatment failure, and CEA response will be assessed.

DETAILED DESCRIPTION:
Approximately 150,000 people are diagnosed with colorectal cancer in the United States each year. Forty to fifty thousand people eventually will develop metastatic colorectal cancer and 40,000 people die annually because of advanced or metastatic colorectal cancer. Cancer patients prefer oral therapy over intravenous therapy as palliative treatment if efficacy regarding response rate and response duration is not compromised. Therefore, development of a completely oral combination therapy that approximates or improves upon the clinical outcomes attained by the reference triple drug therapies should be a research priority. Compared with intravenous 5-fluourouracil/leucovorin as first-line treatment for metastatic colorectal cancer, oral capecitabine has demonstrated similar survival outcomes (approximately 12-13 months), response rates (15-20%), and response durations (4-5 months) in two multi-institutional international randomized phase III trials. Erlotinib (OSI-774, Tarceva) is an orally available inhibitor of human EGFR tyrosine kinase. The epidermal growth factor receptor (EGFR) is overexpressed in a variety of human cancers including colorectal cancer. The principal goal of anticancer treatment with tyrosine kinase inhibitors such as erlotinib is to restore normal cellular growth by interrupting EGFR mediated cell proliferation and malignant The hypothesis of this phase II trial is that the unique mechanisms of action and non-overlapping toxicity profiles of capecitabine (Xeloda) and erlotinib will allow these drugs to be combined into a safe and tolerable regimen with better activity regarding response, response duration, and median survival than capecitabine alone in patients with previously untreated metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have histologically or cytologically confirmed diagnosis of metastatic colorectal adenocarcinoma.
* Patients must be > 18 years old.
* Patients must have a performance status of > 60 on the Karnofsky scale
* Patients must have an expected life expectancy of at least 12 weeks.
* Patients must give written informed consent as per institutional and federal regulatory requirements.
* Patients must have measurable or evaluable disease .
* Patients must have an absolute neutrophil count of > 1,500/mm3 and a platelet count > 100,000/mm3.
* Patients must have adequate liver and renal function defined by a bilirubin of < 2.0 mg/dl and a creatinine of < 1.5 mg/dl, respectively.
* Patients must be able to stay in the general area for the duration of their treatment on this clinical research study.

Exclusion Criteria:

* Prior chemotherapy, treatment with inhibitors of EGFR of any kind, molecularly targeted
* Pregnant or lactating women
* Clinical signs of brain involvement or leptomeningeal disease
* Serious illness or medical conditions
* Congestive heart failure or unstable angina pectoris, uncontrolled hypertension or arrhythmias
* Active infections
* UnstaOphthalmic disorders that might increase the risk for epithelium related complications (bullous keratopathy, aniridia, severe chemical burns, neutrophilic keratitis e.g.)
* GI tract disease resulting in an inability to take oral medication such as uncontrolled inflammatory GI disease (e.g. Crohn's disease, ulcerative colitis) or post surgical malabsorption characterized by uncontrolled diarrhea that results in weight loss and vitamin deficiency orequires IV hyperalimentation (however, use of pancreatic enzyme supplementation is allowed provided that the above criteria are not met).
* Prior invasive malignancies for less 5 years
* Known to be HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To document the antitumor activity of capecitabine in combination with erlotinib in patients with previously untreated metastatic colorectal cancer | Time to tumor progression, time to confirmed response rate, time to treatment failure, .

SECONDARY OUTCOMES:
To determine the qualitative and quantitative toxicity of this combination and sequence of drug administration | Objective response rate, duration of confirmed response rate, CEA response will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kozuch, MD, Principal Investigator — Continuum Cancer Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

REFERENCES:
- [Background] Van Halteren HK, Roumen RM, Coebergh JW, Croiset van Uchelen FA, Keuning JJ, Vreugdenhil G. The impact of 5-FU-based bolus chemotherapy on survival in patients with advanced colorectal cancer. Anticancer Res. 1999 Jul-Aug;19(4C):3447-9. PMID 10629633